CLINICAL TRIAL: NCT00576940
Title: Standard and Immunostimulating Enteral Nutrition in Patients After Extended Gastrointestinal Surgery - A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Standard and Immunostimulating Enteral Nutrition in Surgical Patients
Acronym: ImmuniEteral
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: 1st Department of Surgery, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1st Dept Surg Enteral; Immunoenteral
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-09

CONDITIONS: Gastric Cancer; Pancreatic Cancer
Keywords: enteral nutrition, immunomodulating nutrition
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMEN: 1 (Experimental): Enteral nutrition with immunostimulating diet (IMEN group: formula supplemented with arginine, glutamine, omega-3 fatty acids)
  Interventions: Drug: Reconvan
- SEN (Active Comparator): postoperative enteral nutrition - standard oligopeptic diet
  Interventions: Drug: Peptisorb

INTERVENTIONS:
Drug: Reconvan — isocaloric, immunomodulating entral diet
  Other Names: oligopeptic immunostimulatory diet
  Arms: IMEN: 1
Drug: Peptisorb — isocaloric, isopeptic standard diet
  Other Names: standard enetral diet
  Arms: SEN

SUMMARY:
The aim of the study was to assess the clinical effect of immunomodulating enteral nutrition in patients undergoing resection for gastrointestinal cancer. 196 subjects were randomly assigned into two study groups: standard and immunostimulating. The study failed to demonstrate any clear advantage of routine postoperative immunonutrition in patients undergoing elective upper gastrointestinal surgery

DETAILED DESCRIPTION:
Background&Aim: The administration of immunomodulating enteral diets during postoperative period in patients after major gastrointestinal surgery is intended to reduce the number of postoperative complications and to shorten the hospital stay. The aim of the study was to assess the clinical effect of enteral immunostimulatory nutrition in surgical patients.

Material and Methods: 196 patients undergoing resection for pancreatic and gastric cancer were randomized in double-blind manner to receive early postoperative enteral nutrition with immunostimulating diet (IMEN group: formula supplemented with arginine, glutamine, omega-3 fatty acids) or oligopeptic control (SEN group) between June 2004 and September 2007. Enteral nutrition was started 6 hours after surgery and continued for 7 days, up to target volume of 100 ml/h. All malnourished patients requiring preoperative nutritional therapy were excluded for the study and treated preoperatively. Outcome measures were: number and type of complications, length of hospital stay, mortality, treatment tolerance, liver and kidney function.

Results: One hundred eighty-three patients (91 in SEN, 92 in IMEN group, 69 F, 114 M, mean age 61.2) of 196 initially enrolled were analyzed. There were 2 deaths in both groups. Median postoperative hospital stay was 12.4 days (SD 5.9) in SEN group and 12.9 days (SD 8.0) in IMEN group (p=0.42). Complications were observed in 21 patients (23.1%) in SEN and 23 (25.2%) in IMEN group (p>0.05). 4 (4.4%) patients in SEN group and 4 (4.4%) in IMEN had surgical complications (p>0.05). There were no differences in liver and kidney function, visceral protein concentration and treatment tolerance.

Conclusion: Clinical and laboratory parameters show no benefit of immunomodulating enteral nutrition over standard enteral nutrition in patients after major gastrointestinal surgery as far as complications, hospital stay, mortality and treatment tolerance and safety are considered.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years undergoing subtotal and total gastric resection with lymphadenectomy and pancreatoduodenectomy/ total pancreatectomy with lymphadenectomy, in good general status (Karnofsky > 80, Eastern Cooperative Oncology Group (ECOG) grade 0 or 1); with no confirmed neoplastic dissemination nor distant metastases
* No severe concomitant disease (heart failure, chronic obstructive pulmonary disease [COPD], coronary aortic bypass graft [CABG], etc.)
* No history of known allergies or drug intolerance

Exclusion Criteria:

* Patients with metastatic or unresectable disease
* Pregnant
* In poor general status (Karnofsky <80, Eastern Cooperative Oncology Group (ECOG) > 1)
* With recent history of severe heart, lung, kidney or liver failure
* With history of allergies or drug intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2004-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The ratio of postoperative complications (infectious and surgical) | Postoperative complications

SECONDARY OUTCOMES:
length of hospital stay | length of hospital stay
function of immune system | function of immune system
assessment of liver and kidney function | assessment of liver and kidney function
determination of the treatment tolerance | determination of the treatment tolerance
assessment of visceral protein turnover | assessment of visceral protein turnover

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kulig, MD, PhD, Study Chair — 1st Department of General Surgery
Locations (1):
- 1st Deparment of General Surgery, Krakow, Krkaow, Poland

REFERENCES:
- [Result] Braga M, Gianotti L, Nespoli L, Radaelli G, Di Carlo V. Nutritional approach in malnourished surgical patients: a prospective randomized study. Arch Surg. 2002 Feb;137(2):174-80. doi: 10.1001/archsurg.137.2.174. PMID 11822956
- [Derived] Klek S, Szybinski P, Szczepanek K. Perioperative immunonutrition in surgical cancer patients: a summary of a decade of research. World J Surg. 2014 Apr;38(4):803-12. doi: 10.1007/s00268-013-2323-z. PMID 24178185
- [Derived] Klek S, Sierzega M, Szybinski P, Szczepanek K, Scislo L, Walewska E, Kulig J. The immunomodulating enteral nutrition in malnourished surgical patients - a prospective, randomized, double-blind clinical trial. Clin Nutr. 2011 Jun;30(3):282-8. doi: 10.1016/j.clnu.2010.10.001. Epub 2010 Nov 13. PMID 21074910
- [Derived] Klek S, Kulig J, Sierzega M, Szczepanek K, Szybinski P, Scislo L, Walewska E, Kubisz A, Szczepanik AM. Standard and immunomodulating enteral nutrition in patients after extended gastrointestinal surgery--a prospective, randomized, controlled clinical trial. Clin Nutr. 2008 Aug;27(4):504-12. doi: 10.1016/j.clnu.2008.04.010. Epub 2008 Jun 20. PMID 18571296